CLINICAL TRIAL: NCT06892106
Title: Spinal Cord Injury Rehabilitation: Gut Dysbiosis and Immune Biomarkers As Functional Prognosis Tools and New Therapeutic Targets - a Longitudinal Prospective Cohort Study
Brief Title: Gut Dysbiosis in Spinal Cord Injury Rehabilitation
Acronym: SCIMBIONT
Status: Completed | Type: Observational
Sponsor: Centro Academico Clínico Egas Moniz Health Alliance (Other)
Collaborators: Centro de Reabilitacao do Norte (Other); Unidade Local de Saude de Gaia e Espinho EPE (Other); Aveiro Institute of Biomedicine (iBiMED) (Unknown); Aveiro University (Other)
Responsible Party: Sponsor
Other Study IDs: 246/2019-2
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injury; Gut Dysbiosis; Immune Dysfunction
Keywords: Spinal Cord Injury; Rehabilitation; Gut Microbiota; Immune System; Gut-Immune-CNS Axis
MeSH Terms: conditions — Spinal Cord Injuries; Immune System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Fecal and blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Spinal cord injury patients - A or B AIS classification: Spinal cord injury patients admitted for hospitalization at Centro de Reabilitação do Norte, Unidade Local de Saúde de Gaia / Espinho, E.P.E. with A (complete) or B (sensory incomplete) classification in The American Spinal Injury Association (ASIA) Impairment Scale (AIS)
- Spinal cord injury patients - C or D AIS classification: Spinal cord injury patients admitted for hospitalization at Centro de Reabilitação do Norte, Unidade Local de Saúde de Gaia / Espinho, E.P.E. with C or D (motor incomplete) classification in The American Spinal Injury Association (ASIA) Impairment Scale (AIS)
- Able-bodied controls: Age, gender and body mass index matched control group of participants recruited among able-bodied personnel from Centro de Reabilitação do Norte, Unidade Local de Saúde de Gaia / Espinho, E.P.E. or their relatives, without any known CNS disease

SUMMARY:
The goal of this study is to investigate the role of gut microbiota, and related immune biomarkers and metabolites, in the functional recovery of spinal cord injury patients during the subacute phase. The main question it aims to answer is:

How does gut microbiota dysbiosis impact functional recovery in subacute SCI patients, in a way that future targeted probiotic interventions may improve SCI outcomes?

DETAILED DESCRIPTION:
Background:

Spinal cord injury (SCI) is a devastating condition with no effective cure. Gut dysbiosis and chronic immune dysfunction are common complications that may hinder recovery. This study aims to investigate the role of gut microbiota and related immune biomarkers and metabolites in the functional recovery of SCI patients during the subacute phase. This study hypothesizes that alterations in the gut microbiota and associated immune responses are critical factors influencing recovery trajectories in patients during the subacute phase of SCI.

Therefore, we aim to investigate the intricate relationship between gut microbiota composition, immune biomarkers, and functional outcomes in this population, to develop a probiotic-based therapeutic intervention.

Study Objectives:

* To characterize gut microbiota changes in subacute SCI patients;
* To identify microbiota-based biomarkers for prognosis;
* To correlate gut dysbiosis with systemic inflammation and functional recovery.

Exploratory objective:

- To assess the potential of probiotic-based approaches for therapeutic intervention.

Study Design and Methodology:

This is an observational, longitudinal, prospective cohort study involving 66 patients with subacute SCI (28 patients with A and B classification in ASIA Impairment Scale - AIS and 38 patients with C and D classification in AIS) and 40 able-bodied control participants.

Participant Recruitment and Enrollment:

Participants admitted for hospitalization at Centro de Reabilitação do Norte (CRN)/Unidade Local de Saúde de Gaia e Espinho (ULSGE) were recruited. Inclusion and exclusion criteria were clearly defined to ensure a homogenous study population.

Data Collection:

Clinical data, including neurological assessments, functional outcome measures (e.g., ASIA Impairment Scale, Functional Independence Measure), and demographic information, were collected at three time points:

T1: Admission to the rehabilitation unit (subacute phase). T2: Discharge from the rehabilitation unit. T3: One-year post-injury follow-up. Biological samples, including fecal samples and blood samples, were collected at each time point (T1, T2, and T3).

Laboratory Analyses:

Microbiome Analysis: Fecal samples undergone 16S rRNA gene sequencing to determine gut microbiota composition and diversity.

Immune Biomarker Quantification: Blood samples were analyzed to quantify levels of key inflammatory cytokines, chemokines, and other immune markers.

Metabolite Profiling: Fecal samples, and/or blood samples will be analyzed using metabolomics techniques to identify gut-derived metabolites that may influence recovery.

Statistical Analysis:

Descriptive statistics (means) were calculated for all outcome measures. Data association studies included gut microbiota composition, AIS-based rehabilitation outcomes (percentage improvement), comorbidities (e.g., UTIs), immune biomarkers, and metabolites at T1-T3, with focus on microbiota linked to SCI. Potential confounders (age, gender, injury level, etc.) and biases were accounted for.

Independent group comparisons (e.g., T1 cytokine levels) used t-tests or Mann-Whitney U-tests, while dependent group comparisons (e.g., cytokine changes within AIS groups) used paired t-tests or Wilcoxon tests. ANOVA, multivariate analyses, and generalized linear models (regression, mixed-model repeated measures) assessed inter-group data and associations between gut microbiota changes and functional/immunological outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults (≥18 years) with traumatic spinal cord injury.
* Injury occurred less than 6 months ago (subacute phase).
* Any neurological level of injury (AIS A-D).

Exclusion Criteria:

* Use of probiotics or immunomodulatory drugs in the last month.
* Major gastrointestinal surgery in the last 5 years.
* Active gastrointestinal diseases or other CNS diseases.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients admitted to Centro de Reabilitação do Norte (CRN) / Unidade Local de Saúde de Gaia e Espinho (ULSGE), between 1st of May 2021 and 16th of October 2023, following a traumatic spinal cord injury.
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-10-16 (Actual); Study Completion 2023-10-16 (Actual)

PRIMARY OUTCOMES:
Change in intestinal microbiota | From hospital admission until to one-year post-injury
  Microbiota relative abundance of different taxonomic levels to estimate change in alpha-diversity (diversity within different samples from the same individual) and in beta-diversity (diversity between groups) from hospital admission to 1-year post-injury
Change in functional independence from hospital admission to 1-year post-injury | From hospital admission until to one-year post-injury
  Change in functional independence, as measured by the Spinal Cord Independence Measure, 4th version (SCIM IV) and by Functional Independence Measure (FIM), from hospital admission to 1-year post-injury.
Change in neuromotor impairment from hospital admission to 1-year post-injury | From hospital admission until to one-year post-injury
  Change in the total ASIA Impairment Scale (AIS) motor score from hospital admission to 1-year post-injury.

SECONDARY OUTCOMES:
Change in bowel function from hospital admission to 1-year post-injury | From hospital admission until to one-year post-injury
  Change in bowel function, as measured by the Neurogenic Bowel Dysfunction (NBD) Score, from hospital admission to 1-year post-injury.
Change in immunological and inflammation biomarkers | From hospital admission until to one-year post-injury
  Change in immunologic and inflammatory serum biomarkers (interleukins, cytokines), measured via ELISA techniques -TNF-alfa, IL-1beta, IL-6, IL-8 and IL-10, IL-1alfa and cytokine MIP2 - from hospital admission to 1-year post-injury.
Change in gut microbiota-produced metabolites | From hospital admission until to one-year post-injury
  Change in gut microbiota-produced metabolites, measured by Nuclear Magnetic Resonance (NMR) and Liquid Chromatography-Mass Spectrometry (LC-MS/MS), from hospital admission to 1-year post-injury

CONTACTS AND LOCATIONS:
Overall Officials: Maria Ribeiro da Cunha, PhD, Principal Investigator — Centro de Reabilitação do Norte (CRN) / Unidade Local de Saúde Gaia e Espinho (ULSGE)); Sandra Vieira, Study Director — Institute of Biomedicine - Aveiro University (iBiMED-UA)
Locations (1):
- Centro de Reabilitação do Norte (CRN) / Unidade Local de Saúde Gaia e Espinho (ULSGE), Vila Nova de Gaia, Porto District, Portugal

IPD SHARING:
Plan to Share IPD: Undecided